CLINICAL TRIAL: NCT05264025
Title: Fexofenadine as Adjunct to Standard Rheumatoid Therapy in Patients With Active Rheumatoid
Brief Title: Fexofenadine in Patients With Active Rheumatoid Arthritis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, engy wahsh, lecturer of clinical pharmacy, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FMBSUREC/08052022/Ismaeel
Record Dates: First submitted 2022-01-10; First posted 2022-03-03 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — fexofenadine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fexo group (Active Comparator)
  Interventions: Drug: Fexofenadine
- Placepo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fexofenadine — tablet
  Arms: Fexo group
Drug: Placebo — tablet
  Arms: Placepo

SUMMARY:
Rheumatoid arthritis (RA) is an inflammatory autoimmune polyarthritis affecting ∼1% of the world population, resulting in the loss of joint function and progressive structural damage in affected joints. Fexofenadine has been widely used to treat various allergic diseases, like allergic rhinitis, conjunctivitis and chronic idiopathic urticaria. the molecular mechanisms underlying fexofenadine mediated inhibition of TNF-α signalling

ELIGIBILITY:
Inclusion Criteria

* Moderate to severe RA (disease activity score-28 joints: DAS-28 > 3.2) were recruited.
* Age between 18 - 60 years having active disease according to the diagnosis of an experienced rheumatologist, being under treatment with disease-modifying anti-rheumatic drugs (DMARDs), not receiving cytokine inhibitors
* Signing informed consent and willingness of the participant to accept randomization to any assigned treatment arm.

Exclusion Criteria:

* History of biological DMARDS.
* History/presence of acute heart disease, liver and kidney diseases, COPD
* Intolerance or allergy to fexofenadine or methotrexate
* Alcohol abuse
* Any changes in using medication (changing the dosage or type of medicines
* Receive hormone replacement therapy, warfarin, and other anticoagulants

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
ACR 20% | at baseline
  improvement criteria (ACR20) response rate based on the count of tender/swollen joints,
ACR 20% | at week 12
  improvement criteria (ACR20) response rate based on the count of tender/swollen joints,
(HAQDI) | at baseline
  HAQ-DI (Health Assessment Score- Disability index), in which patients are asked to rate their capacity to perform 20 activities of daily living (ADL). Scoring within each section is from 0 (without any difficulty) to 3 (unable to do). For each section the score given to that section is the worst score within the section
(HAQDI) | at week 12
  HAQ-DI (Health Assessment Score- Disability index), in which patients are asked to rate their capacity to perform 20 activities of daily living (ADL). Scoring within each section is from 0 (without any difficulty) to 3 (unable to do). For each section the score given to that section is the worst score within the section
CRP | at baseline
  the level of CRP
CRP | at week 12
  the level of CRP

SECONDARY OUTCOMES:
TNF-α | at baseline and at week 12
  Serum level Tumor necrosis factor- alpha (TNF-α)
IL6 | at baseline and at week 12
  Serum level of IL6

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Beni-Suef Hospital, Banī Suwayf
  - Faculty of Medicine - Beni Suef Hospital, Banī Suwayf

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP